CLINICAL TRIAL: NCT00815399
Title: Effect of Pioglitazone Compared With Metformin on Endothelial Microparticles in Type 2 Diabetes. A Randomized Trial
Brief Title: Pioglitazone Versus Metformin in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Dario Giugliano, Prof of Endocrinology and Metabolism, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMD/2007/10
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pioglitazone
- 2 (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Pioglitazone — 15-45 mg/die
  Arms: 1
Drug: Metformin — 500-2000 mg/die
  Arms: 2

SUMMARY:
Type 2 diabetes is an epidemic. Its long-term consequences translate into enormous human suffering and economic costs; however, much of the morbidity associated with long-term microvascular and neuropathic complications can be substantially reduced by interventions that achieve glucose levels close to the nondiabetic range. However, none of the recent intervention studies has demonstrated a benefit of intensive glycemic control on their primary CVD outcomes.

The investigators report the findings of a long-term randomized and comparator-controlled clinical trial conducted in patients with newly-diagnosed type 2 diabetes. The investigators compared the effect of pioglitazone with that of metformin on circulating endothelial cell-derived submicroscopic membranous vesicles, termed microparticles: because of their putative role in inflammatory processes and their ability to directly affect endothelial functions, they are gaining increasing popularity as a surrogate marker of cardiovascular outlook. Metformin was chosen as a comparator because the American Diabetes Association recommendations suggest to start therapy in newly-diagnosed type 2 diabetic subjects combining a drug (metformin) with lifestyle changes. Moreover, the mechanism of action of pioglitazone is distinct from that of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 30-75 years, with newly-diagnosed type 2 diabetes (according to the ADA criteria) and never treated with antihyperglycemic drugs, were selected for the study. Inclusion criteria also included a body mass index (BMI) >25 kg/m2, and HbA1c level <10%.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Any investigational drug within the previous 3 months
* Use of agents affecting glycemic control (systemic glucocorticoids, and weight-loss drugs)
* Presence of any clinically relevant somatic or mental diseases that anticipated poor adherence to diet regimens
* To minimize the likelihood of including subjects with late-onset type 1 diabetes, candidates with a positive test for anti-GAD antibody or with fasting plasma C-peptide less than 0.76 ng/L (<0.25 pmol/L) were excluded
* Also excluded were patients with abnormal laboratory tests, including liver enzymes (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase) greater than 3 times the upper limit of normal, and serum creatinine greater than 123.8 μmol/L (1.4 mg/dL).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-10; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Circulating Endothelial microparticles | six months

SECONDARY OUTCOMES:
Glucose profile, lipid profile, hemoglobin A1c, carotid intima-media thickness | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatrics and Metabolic Diseases, Naples, Italy

REFERENCES:
- [Background] Mazzone T, Meyer PM, Feinstein SB, Davidson MH, Kondos GT, D'Agostino RB Sr, Perez A, Provost JC, Haffner SM. Effect of pioglitazone compared with glimepiride on carotid intima-media thickness in type 2 diabetes: a randomized trial. JAMA. 2006 Dec 6;296(21):2572-81. doi: 10.1001/jama.296.21.joc60158. Epub 2006 Nov 13. PMID 17101640